CLINICAL TRIAL: NCT03855826
Title: Evaluation of the Efficacy and Safety of Nifekalant Hydrochloride (NIF) Injection in the Treatment of Ventricular Tachycardia and Ventricular Fibrillation. A Multicenter, Randomized, Controlled, Open-label, Clinical Trial.
Brief Title: Evaluation of the Efficacy and Safety of Nifekalant Hydrochloride (NIF) Injection.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTFS01
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation | interventions — nifekalant; Injections; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nifekalant Hydrochloride (Experimental): Nifekalant hydrochloride (50mg) should be dissolved into a 50ml dilution solution (0.9% sodium chloride injection or 5% glucose injection), and configured as 1mg/ml solution of nificaine hydrochloride. The dosage should be taken as needed. The diluted solution should be used within 24 hours. The amount of fluid per hour should not exceed 50ml when intravenously infused. It is recommended to use intravenous pump.
  Interventions: Drug: Nifekalant hydrochloride
- Amiodarone (Active Comparator): The concentration of more than 2 ampoule amiodarone injection in 500 ml (only isotonic grape solution) is suitable. Amiodarone should be administered as far as possible via the central venous route (administered separately).
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Nifekalant hydrochloride — Both groups were given conventional treatment except for arrhythmia drugs.Only nyficarine hydrochloride or amiodarone hydrochloride could be used according to random results, and the antiarrhythmic drugs should be replaced according to the protocol rules.
  Other Names: Nifekalant Hydrochloride for Injection
  Arms: Nifekalant Hydrochloride
Drug: Amiodarone — Both groups were given conventional treatment except for arrhythmia drugs.Only nyficarine hydrochloride or amiodarone hydrochloride could be used according to random results, and the antiarrhythmic drugs should be replaced according to the protocol rules.
  Other Names: Amiodarone hydrochloride
  Arms: Amiodarone

SUMMARY:
Efficacy and safety evaluation of amiodarone and Nifekalant hydrochloride(NIF) for the treatment of ventricular tachycardia and ventricular fibrillation.

DETAILED DESCRIPTION:
After patients are hospitalized, they will be treated as usual in addition to antiarrhythmic drugs. DC will be performed again according to normal procedures for patients who were ineffective. Arrhythmia drugs can only be used with nifekalant or amiodarone at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent ventricular tachycardia or ventricular fibrillation who have a combined physical heart disease, or who have a conventional drug ineffective or persistent idiopathic ventricular tachycardia with amiodarone indications;
* Age ≥ 18 years old, gender is not limited.

Exclusion Criteria:

* Patients with prolonged ventricular tachycardia with QT interval and patients with QTc interval of more than 500 ms before administration;
* Patients with torsades de pointes (Tdp);
* Patients with Brugada syndrome;
* Patients with severe atrioventricular block and without pacing protection;
* Patients with hypertrophic cardiomyopathy (HCM) with ventricular septal thickness or (and) left ventricular wall ≥ 15 mm;
* Pregnant or lactating women;
* Patients who are not suitable for the study, considered by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
The rate of efficacy | 24 hours after administration.
  Efficacy of drugs in each group within 24 hours after administration.

SECONDARY OUTCOMES:
The efficiency rate without adjusting the drug dose | 24 hours after administration.
  number of patients who no longer relapse after using the drug / total number of patients in the group × 100%
Number of electrical cardioversion used during the treatment | 24 hours after administration.
  Number of electrical cardioversion
The success rate of DC in patients with first invalid cardioversion in the two groups | 24 hours after administration.
  Number of patients ewith valid DC after the first invalid DC / Total number of patients with first invalid DC in this group × 100%
The average time from the start of administration to the last VT/VF no longer occurs | 24 hours after administration.
  Patients who changed drugs will not be included statistics on this indicator.
LVEF | Before administration, and 24h to 72h after the start of administration.
  Echocardiography
Survival rate | 30 days after administration.
  Survival rate of the two groups of patients
Number of ventricular tachycardia/ventricular fibrillation episodes | Within 72 hours after drug administration.
  Number of ventricular tachycardia/ventricular fibrillation episodes .
The number of patients who need to continue the intravenous research drug after 24 hours in the two groups | 24 hours after the start of the adminstration.
  The number of patients who need to continue the intravenous research drug after 24 hours in the two groups
The effective rate of the drug in each group within 72 hours after administration | 72 hours after administration.
  The effective rate of the drug in each group within 72 hours after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Ya Han, Principal Investigator — Shenyang Military Region General Hospital
Locations (1):
- Shenyang Military Region General Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided